CLINICAL TRIAL: NCT00845221
Title: Glivec in Pediatric Chronic Myeloid Leukemia (CML)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Docteur Frédéric MILLOT/principal investigator, CHU DE POITIERS
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: GLIVEC PHASE IV
Record Dates: First submitted 2009-02-16; First posted 2009-02-18 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-10

CONDITIONS: Chronic Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Imatinib Mesylate

ARMS (1):
- Imatinib (Experimental)
  Interventions: Drug: Imatinib mesylate 100 mg (Glivec)

INTERVENTIONS:
Drug: Imatinib mesylate 100 mg (Glivec) — 260 mg/m2/day tablets

SUMMARY:
It is a phase 4 study, not randomised and multicentric. Within 2 months after the diagnosis, the patients daily receive imatinib by oral way during at least 1 year (260mg/m² once a day), i.e. until the cytogenetic analysis.

Beyond 1 year of treatment, if a haematological relapse or a loss of the cytogenetic response is observed, the nature of the treatment suggested to the patient is left with the appreciation of the investigator.

Later on, discontinuation of imatinib is discussed if a molecular remission (negative RT-PCR) is obtained and maintained for at least 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Old < 18 years, male or female.
* Chronic myeloid leukaemia confirmed on the cytogenetic level by the presence of the translocation t(9; 22) (q34; q11) or by the presence of transcript BCR-ABL in the event of absence of description of the translocation t(9; 22) (q34; q11).
* Chronic phase of a chronic myeloid leukaemia
* Absence of extra-medullary disease (except for a hepatomegaly and/or of a splenomegaly).
* Absence of any former treatment of chronic myeloid leukaemia except for hydroxyurea.
* Stop of hydroxyurea at least week before the beginning of the imatinib mesylate.
* Diagnosis of chronic myeloid leukaemia in chronic phase recent (less than 2 months).
* Score of Lansky ≥ 60.
* Effective contraception among patients in age to procreate.
* Written voluntary informed consent of the two parents or the legal guardian.

Exclusion Criteria:

* Patients with grade 3 / 4 cardiac disease.
* Pathology cardiac, pulmonary, hepatic, renal or neurological of grade > 2 (WHO).
* Participation in a clinical trial in the 28 days preceding the beginning by the treatment.
* Impossible Follow-up during at least 2 years, patient not compliant.
* Expectant mother or nursing.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Actual)
Dates: Start 2004-07; Primary Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CHU Amiens, Amiens
  - Hôpital La Timone - CHU de Marseille, Marseille
  - Hôpital de Brabois - CHU de Nancy, Vendoeuvre Les Nancy

REFERENCES:
- [Derived] Millot F, Guilhot J, Baruchel A, Petit A, Bertrand Y, Mazingue F, Lutz P, Verite C, Berthou C, Galambrun C, Sirvent N, Yakouben K, Schmitt C, Gandemer V, Reguerre Y, Couillault G, Mechinaud F, Cayuela JM. Impact of early molecular response in children with chronic myeloid leukemia treated in the French Glivec phase 4 study. Blood. 2014 Oct 9;124(15):2408-10. doi: 10.1182/blood-2014-05-578567. Epub 2014 Aug 28. PMID 25170123
- [Derived] Millot F, Baruchel A, Guilhot J, Petit A, Leblanc T, Bertrand Y, Mazingue F, Lutz P, Verite C, Berthou C, Galambrun C, Bernard F, Yacouben K, Bordigoni P, Edan C, Reguerre Y, Couillault G, Mechinaud F, Cayuela JM, Guilhot F. Imatinib is effective in children with previously untreated chronic myelogenous leukemia in early chronic phase: results of the French national phase IV trial. J Clin Oncol. 2011 Jul 10;29(20):2827-32. doi: 10.1200/JCO.2010.32.7114. Epub 2011 Jun 13. PMID 21670449